CLINICAL TRIAL: NCT04877769
Title: A Phase 1, Open-label, Randomized Study in Healthy Subjects to Assess the Bronchopulmonary Pharmacokinetics, Safety and Tolerability of AT-527, a Potential Treatment for COVID-19
Brief Title: Bronchopulmonary PK of AT-527 (R07496998)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT-03A-007
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2021-04

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — AT-511

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- AT-527 Group A (Experimental): n=8
  Interventions: Drug: AT-527
- AT-527 Group B (Experimental): n=8
  Interventions: Drug: AT-527
- AT-527 Group C (Experimental): n=8
  Interventions: Drug: AT-527

INTERVENTIONS:
Drug: AT-527 — administered twice daily (BID) for 2.5 days (5 doses in total)
  Other Names: RO7496998

SUMMARY:
This study will assess the safety, tolerability and bronchopulmonary pharmacokinetics (PK) of AT-527 (R07496998)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must agree to use birth control, as required by the protocol.
* Females must have a negative pregnancy test at Screening and prior to dosing
* Minimum body weight of 50 kg and body mass index (BMI) of 18-29 kg/m2
* Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV or SARS-CoV-2
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Concomitant use of prescription medications, or systemic over-the-counter medications
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Concentrations of AT-527 in epithelial lining fluid | 4-5 hours after last dose and 11-12 hours after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, London, United Kingdom